CLINICAL TRIAL: NCT01393392
Title: Developing a Smoking Cessation Intervention for Methadone Maintained Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nina A. Copperman, Psy. D., Associate Professor of Psychiatry, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23DA025049 (NIH); K23DA025049 (NIH)
Record Dates: First submitted 2011-06-27; First posted 2011-07-13 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Nicotine Dependence; Opiate Dependence
Keywords: smoking cessation; methadone treatment; nicotine addiction; drug treatment; drug addiction; tobacco dependence
MeSH Terms: conditions — Tobacco Use Disorder; Opioid-Related Disorders; Smoking Cessation; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive, tailored intervention (Experimental): Participants in the intensive intervention condition will receive eight individual counseling sessions, with a smoking cessation counselor, over three months. Each session will last approximately 45 minutes and occur in the methadone clinic. Participant treatment needs will be assessed during the first session and the intervention will be tailored to the participants' needs. Prior to quitting participants will receive nicotine replacement patches and lozenges and instructions on how to use them.
  Interventions: Behavioral: Intensive, tailored intervention
- Control Intervention (Active Comparator): Participants randomized to the control intervention will receive a referral to the NJ Quitline (a telephone smoking cessation counseling service). Participants will receive a brochure and information about the referral. Study staff will contact the NJ Quitline for control participants, and a counselor from the Quitline will call control participants.
  Interventions: Behavioral: NJ Quitline Referral

INTERVENTIONS:
Behavioral: Intensive, tailored intervention — Eight, 45 minute counseling sessions, tailored to the individual and based on the Information-Motivation-Behavioral Skills model of behavior change. Incorporates motivational interviewing, education, cognitive-behavioral skills training. 12 week course of nicotine replacement patches provided. Nicotine lozenges also provided.
  Other Names: Smokers in Methadone Treatment Intervention; IMB Model Based Smoking Cessation Intervention
  Arms: Intensive, tailored intervention
Behavioral: NJ Quitline Referral — Participants will receive a facilitated referral to the NJ Quitline (i.e. fax to quit).
  Other Names: Standard of Care Smoking Cessation Intervention; General Population Smoking Cessation Intervention
  Arms: Control Intervention

SUMMARY:
The purpose of this study is to pilot and evaluate, in a randomized controlled trial, the immediate and long-term effects of a newly developed, tailored, intensive smoking cessation intervention among methadone maintained smokers and compared to a control condition (facilitated referral to the NJ Quitline). The newly developed intervention is evidence based, addresses the unique needs of methadone maintained smokers, is intensive, can be tailored to the individual, and builds on the strengths as well as addresses the gaps in previous treatments for methadone maintained smokers.

The investigators hypothesize that: (1) three months and six months after beginning treatment, those in the tailored intervention condition will be more likely to be abstinent from smoking than those in the control intervention condition (primary outcome); (2) there will be a greater relapse rate in the control intervention condition between the three and six month follow-up points than in the tailored intervention condition; (3) three and six months after beginning treatment, those in the tailored intervention condition will have better secondary smoking related outcomes (smoked fewer cigarettes per day in the past week, be more ready to quit, have greater self-efficacy for quitting, experience less nicotine dependence, and be more likely to have made a quit attempt) than those in the control intervention condition; (4) three and six months after beginning treatment, those in the tailored intervention condition will have better utilization of and adherence to smoking cessation pharmacotherapy, better mental and physical health, less perceived stress, greater social support, less drug and alcohol use, and greater involvement in drug and alcohol treatment than those in the control intervention condition; and (5) the newly created tailored intervention will be feasible and acceptable. .

DETAILED DESCRIPTION:
Most individuals in methadone maintenance treatment are tobacco smokers. Also, people in methadone treatment are more likely to experience the health issues related to smoking than the general population. Yet, research has found that smokers receiving methadone treatment are interested in quitting and receiving tobacco cessation treatment, and people in drug treatment who quit smoking are less likely to use drugs.

To better help methadone maintained smokers quit smoking and prevent them from starting smoking again, we want to evaluate the effects of a new smoking cessation counseling intervention, designed for methadone maintained smokers as compared to a smoking cessation counseling intervention used with the general population.

Eligible participants will:

* Be English speaking (i.e., able to participate in counseling sessions in English and to complete study interviews in English);
* Be enrolled in methadone treatment for at least three months;
* Be able to give informed consent;
* Be willing and able to participate in all study activities;
* Not have taken smoking cessation related medication or participated in smoking cessation counseling in the past six months;
* Have smoked at least 100 cigarettes during their lifetime and currently smoke every day or most days;
* Not currently be pregnant or breastfeeding or plan on getting pregnant or breastfeeding during the next six months;
* Have access to a working telephone; and,
* Be interested in participating in a smoking cessation intervention and quitting smoking within the next six months.

Participants will be randomly assigned to receive either a smoking cessation intervention tailored for methadone maintained smokers or a referral to a smoking cessation program available to the general population (NJ Quitline). Participants assigned to receive the tailored intervention, will participate in approximately eight individual counseling sessions, with a smoking cessation counselor, over three months. Each session will last approximately 45 minutes and occur in the participant's methadone clinic. Treatment needs will be assessed during the first session and the intervention will be tailored to participants' needs. Prior to quitting participants will receive nicotine replacement patches and lozenges and instructions on how to use them.

Study staff will contact the NJ Quitline for participants assigned to the control condition, and a counselor from the Quitline will call them.

Regardless of treatment assignment, participants will be asked to provide a urine sample for a drug test and pregnancy test (for women) and complete an interview, using a computer or face-to-face, before beginning treatment or receiving the NJ Quitline referral and three months and six months after study enrollment.Each interview will take approximately 45 minutes to one hour to complete.

Participants will receive a $20 gift card for completing each research visit (i.e., computer or face-to-face interview), but will not be reimbursed for counseling visits.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in methadone treatment for at least three months
* Able to give informed consent
* Willing and able to participate in all study activities
* Smoked at least 100 cigarettes during their lifetime
* Currently smoke every day or most days
* Has access to a working telephone
* Interested in participating in a smoking cessation intervention and quitting smoking within the next six months

Exclusion Criteria:

* Unable to speak English fluently
* Took smoking cessation related medication or participated in smoking cessation counseling in the past three months
* Pregnant or breastfeeding or planning on becoming pregnant or breastfeeding during the next six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Cooperman, Psy.D., Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive, Tailored Intervention | Control Intervention
Started | 44 | 43
Completed | 33 | 24
Not Completed | 11 | 19

BASELINE CHARACTERISTICS:
Population: Intensive, tailored intervention: n=41 included in analyses (n=3 did not receive allocated intervention 1 dropped from methadone program before any sessions and two never came to sessions or research visits)
  Control Intervention:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive, Tailored Intervention | Control Intervention | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (11) | 42 (10) | 43 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 32 | 34 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 31 | 31 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Seven-day Point Prevalence Smoking Abstinence
Description: Self-reported not smoking "even a puff" within the previous seven days, and exhaled carbon monoxide reading of <8 parts per million.
Time Frame: during the previous seven days at three months post baseline
Population: Three individuals randomized to the intensive, tailored intervention group did not attend any intervention sessions, and one participant in the control condition passed away; these individuals were not included in the analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Tailored Intervention | Control Intervention
Number analyzed (Participants) | 41 | 42
Participants | 3 | 0

2. Secondary Outcome: Median Number of Cigarettes Participants Smoked Per Day During the Past Week
Description: Self-reported, median number of cigarettes per day during the previous seven days
Time Frame: during the previous seven days at three months post baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cigarettes
Arm/Group | Intensive, Tailored Intervention | Control Intervention
Number analyzed (Participants) | 41 | 42
cigarettes | 6 [4 to 15] | 10 [5 to 20]

3. Secondary Outcome: Number of Participants Who Experienced Any Quit Attempts Since Baseline
Description: Self-reported, smoke free for 24 hours or more since baseline (yes/no)
Time Frame: During the period between baseline and three months post enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Tailored Intervention | Control Intervention
Number analyzed (Participants) | 41 | 42
Participants | 21 | 14

4. Secondary Outcome: Number of Participants Who Experienced Seven-day Point Prevalence of Smoking Abstinence
Description: as for outcome 1
Time Frame: during the previous seven days at six months post baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Tailored Intervention | Control Intervention
Number analyzed (Participants) | 41 | 42
Participants | 1 | 0

5. Secondary Outcome: Median Number of Cigarettes Smoked Per Day During the Past Week
Description: Self-reported, median number of cigarettes per day during the previous seven days
Time Frame: during the previous seven days at six months post baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cigarettes
Arm/Group | Intensive, Tailored Intervention | Control Intervention
Number analyzed (Participants) | 41 | 42
cigarettes | 8 [4 to 14] | 10 [6 to 20]

6. Secondary Outcome: Number of Participants Who Experienced Any Quit Attempts Since Enrollment
Description: Self-reported, smoke free for 24 hours or more since baseline (yes/no)
Time Frame: during the period between baseline and six months post-enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Tailored Intervention | Control Intervention
Number analyzed (Participants) | 41 | 42
Participants | 23 | 17

ADVERSE EVENTS:
Time Frame: 2.5 years
Description: AEs assessed at each counseling and research visit.
Arm/Group | Intensive, Tailored Intervention | Control Intervention
All-Cause Mortality (participants affected / at risk) | 0/44 | 1/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/43
Other Adverse Events (participants affected / at risk) | 20/44 | 1/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive, Tailored Intervention (N=44) | Control Intervention (N=43)
Death (Renal and urinary disorders) | 0 (0) | 1 (1) — Death related to pre-existing kidney disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive, Tailored Intervention (N=44) | Control Intervention (N=43)
cough up blood (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
leg pain (General disorders) | 2 (2) | 0 (0)
nausea (General disorders) | 2 (2) | 0 (0)
insomnia (General disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 5 (5) | 0 (0)
increased alcohol use (General disorders) | 1 (1) | 0 (0)
itching/irritation at patch site (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
jittery/agitated/irritable (General disorders) | 4 (4) | 0 (0)
tooth infection (Infections and infestations) | 1 (1) | 0 (0)
headache (General disorders) | 3 (3) | 0 (0)
vivid dreams (General disorders) | 2 (2) | 0 (0)
hemorrhoids (General disorders) | 1 (1) | 0 (0)
chest discomfort/pain (General disorders) | 2 (2) | 0 (0)
increased appetite (General disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Extremely high expired carbon monoxide level (General disorders) | 1 (1) | 0 (0)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sores on tongue (General disorders) | 1 (1) | 0 (0)
suicidal ideation (Psychiatric disorders) | 2 (2) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
insomnia/restless sleep (General disorders) | 2 (2) | 0 (0)
vertigo (General disorders) | 2 (2) | 0 (0)
anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
appendicitis (General disorders) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 1 (1) | 0 (0)
cough (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No